CLINICAL TRIAL: NCT04608045
Title: A Phase 1, First-in-Human, Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics Study of CPX-POM in Patients With Advanced Solid Tumors
Brief Title: Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics Study of CPX-POM in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CicloMed LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPX-POM-01-001EXP
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-POM, 900 mg/m2 by 20 minute IV infusion (Experimental)
  Interventions: Drug: CPX-POM

INTERVENTIONS:
Drug: CPX-POM — CPX-POM

SUMMARY:
The expansion study was a Phase I, multicenter, open label feasibility trial to characterize the pharmacologic activity of IV CPX-POM in bladder tumor tissues obtained from patients with MIBC (Stage ≥T2, N0-N1, M0) who were scheduled for RC with bilateral (standard or extended) pelvic lymph node dissection (PLND).

The Dose Escalation study was a Phase I, multicenter, open label, dose escalation study to evaluate the DLTs and MTD and to determine the recommended Phase 2 dose (RP2D) of CPX-POM administered IV in patients with any histologically- or cytologically-confirmed solid tumor type and was completed.

DETAILED DESCRIPTION:
The expansion cohort of this study was conducted at up to 3 study sites. It was an open-label feasibility trial to characterize the pharmacologic activity of IV CPX-POM in bladder tumor tissues obtained from patients with MIBC (Stage ≥T2, N0-N1, M0) who were scheduled for RC with bilateral (standard or extended) pelvic lymph node dissection (PLND). Both cisplatin eligible and chemotherapy eligible MIBC patients scheduled for RC were eligible to participate. Neoadjuvant treatment with CPX-POM, whether alone or in combination with gemcitabine +cisplatin, started within 8 weeks of transurethral resection of the bladder tumor (TURBT) that showed muscularis propria invasion.

Nine patients, four cisplatin-ineligible, and five chemotherapy-eligible patients, were enrolled. Patients who are cisplatin-ineligible were treated with two 21-day treatment cycles of CPX-POM alone (Cycle 1, Days 1-5 treatment, rest days 6-21; Cycle 2, Days 22-26 treatment, rest days 27-43) before a planned RC. Chemotherapy-eligible patients received neoadjuvant chemotherapy (gemcitabine + cisplatin in three 21-day treatment cycles) in combination with three 21-day treatment cycles of CPX-POM (Cycle 1, Days 1-5 treatment, rest days 6-21; Cycle 2, Days 22-26 treatment, rest days 27-42; Cycle 3, Days 43-47, rest days 48-63), i.e. concurrently with the prescribed chemotherapy. The cisplatin + gemcitabine dosing regimen for chemotherapy-eligible patients in the Expansion Cohort was administered per the institution's standard of care. After each infusion of CPX-POM at the RP2D of 900 mg/m2,, patients remained in the clinic for at least a 1-hour observation period. On Day 1 of Cycle 1, single blood and clean catch urine samples were collected prior to the first CPX-POM infusion. On Day 5 of Cycle 1, serial blood and complete urine samples were collected over 24 hours following the fifth, once daily CPX-POM RP2D dose of 900 mg/m2 infused over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged ≥18 years.
2. Patient provided signed and dated informed consent prior to initiation of any study procedures.
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
4. Patient has a predicted life expectancy of ≥3 months.
5. Patient has a GFR of ≥30 mL/min/1.73 m^2.
6. Patient has adequate hepatic function, as evidenced by a total bilirubin ≤1.5 × ULN, aspartate transaminase (AST), and /or alanine transaminase (ALT) ≤3 × ULN or ≤5 ×ULN, if due to liver involvement by tumor.
7. Patient has adequate bone marrow function, as evidenced by hemoglobin ≥9.0 g/dL in the absence of transfusion within the previous 72 hours, platelet count ≥100×10^9cells/L, and absolute neutrophil count (ANC) ≥1.5×10^9 cells/L.
8. Patient has no significant ischemic heart disease or myocardial infarction (MI) within 6 months before the first dose of CPX-POM and currently has adequate cardiac function, as evidenced by a left ventricular ejection fraction of >50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO); and corrected QT interval (QTc) <470 msec by Fridericia (QTcF). The eligibility of patients with ventricular pacemakers for whom the QT interval may not be accurately measurable will be determined on a case by-case basis by the Sponsor in consultation with the Medical Monitor.
9. Patient and his/her partner agree to use adequate contraception after providing written informed consent through 3 months after the last dose of CPX-POM, as follows:

   1. For women: Negative pregnancy test during Screening and at Day 1 of each treatment cycle and compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile or postmenopausal.
   2. For men: Compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile. Men whose sexual partners are of child-bearing potential must agree to use 2 methods of contraception prior to study entry, during the study, and for 3 months after the treatment period.
10. Patient is willing and able to participate in the study and comply with all study requirements.
11. Patients must have histologically confirmed MIBC (≥T2, N0-N1, M0 per AJCC) pure or mixed histology urothelial carcinoma. Clinical node-positive (N1) patients are eligible provided the lymph nodes (LNs) are confined to the true pelvis and are within the planned surgical LN dissection template.
12. The initial TURBT that showed muscularis propria invasion should be within 8 weeks prior to beginning study therapy, when feasible. There must be adequate evaluable tumor burden in the tissue blocks (from initial or repeat TURBT with highest tumor content) to allow for analysis as determined by the local site pathologist.
13. Patients must be ineligible for cisplatin-based chemotherapy due to any of the following:

    1. Creatinine clearance(CrCl) <60 mL/min with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
    2. Hearing impaired ≥ Grade 2 by CTCAE criteria
    3. Neuropathy ≥ Grade 2 by CTCAE criteria
    4. Heart failure New York Heart Association (NYHA) ≥ III

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in the Expansion Cohort.

1. Baseline GFR <30 mL/min/1.73 m^2.
2. Women must not be pregnant or breastfeeding since we do not know the effects of CPX-POM on the fetus or breastfeeding child.
3. Patients may not have concurrent upper urinary tract (i.e. ureter, renal pelvis) invasive urothelial carcinoma. Patients with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.
4. Patients may not have another malignancy that could interfere with the evaluation of safety or efficacy of the study drugs. Patients with a prior malignancy will be allowed without study chair approval in the following circumstances:

   1. Not currently active and diagnosed at least 3 years prior to the date of registration.
   2. Non-invasive diseases such as low risk cervical cancer or any cancer in situ.
   3. Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy), and in which no chemotherapy was indicated.( (e.g. low/ intermediate risk prostate cancer, etc.).
5. Patients may not have undergone major surgery with the exception of TURBT (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury or specific anti-cancer treatment ≤ 4 weeks prior to starting study drug, or patients who have had percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury.
6. Patients must not have clinically significant cardiac disease.
7. Patients may not have chronic active liver disease or evidence of acute or chronic Hepatitis B Virus (HBV) or Hepatitis C (HCV).
8. Patients may not have known diagnosis of human immunodeficiency virus (HIV) infection. Testing is not required in absence of clinical suspicion.
9. Patients may not have known diagnosis of any condition (e.g. post hematopoietic or solid organ transplant, pneumonitis, inflammatory bowel disease, etc.) that requires chronic immunosuppressive therapy. Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted.
10. Patients with any serious and/or uncontrolled concurrent medical conditions (e.g.., active or uncontrolled infection, uncontrolled diabetes) or psychiatric illness that could, in the investigator's opinion, cause unacceptable safety risks or potentially interfere with the completion of the treatment according to the protocol are not eligible.
11. Patients may not have any live viral vaccine used for prevention of infectious diseases within 4 weeks prior to study drug(s).
12. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-19 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Taylor III, MD, MSc, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weir SJ, Dandawate P, Standing D, Bhattacharyya S, Ramamoorthy P, Rangarajan P, Wood R, Brinker AE, Woolbright BL, Tanol M, Ham T, McCulloch W, Dalton M, Reed GA, Baltezor MJ, Jensen RA, Taylor JA 3rd, Anant S. Fosciclopirox suppresses growth of high-grade urothelial cancer by targeting the gamma-secretase complex. Cell Death Dis. 2021 May 31;12(6):562. doi: 10.1038/s41419-021-03836-z. PMID 34059639
- See also: CPX-POM-01-001 study — https://clinicaltrials.gov/ct2/show/NCT03348514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CPX-POM-001EXP (NCT04608045) was submitted to and approved by FDA as a protocol amendment to CPX-POM-001 (dose escalation study, NCT03348514), the Phase 1 Dose Escalation Study.
  The dosage regimen was determined to be the Recommended Phase 2 Dose (RP2D) defined by the CPX-POM-001 Dose Escalation Study (NCT03348514) conducted in advanced solid tumor patients. The nine patients enrolled in CPX-POM-001EXP (NCT04608045) received one dosage regimen of 900 mg/m^2 via a 20-minute infusion.
Pre-assignment Details: CPX-POM-001EXP was conducted in muscle-invasive bladder cancer (MIBC) patients scheduled for cystectomy. MIBC, cisplatin-ineligible MIBC and cisplatin-eligible MIBC patients received fosciclopirox for 2 or 3, 21-day treatment, fosciclopirox alone prior to cystectomy for 2, 21-day treatment cycles or fosciclopirox for 3, 21-day treatment cycles in combination with standard-of-care gemcitabine and cisplatin prior to cystectomy. The dosage regimen was administered in a neoadjuvant setting.
Groups:
- CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion: CPX-POM: CPX-POM
Period: Overall Study
Arm/Group | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion
Started | 9
Completed | 8
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Determine Disease Response Following 2 or 3 CPX-POM Treatment Cycles by Assessing the Complete and Partial Pathologic Response Rate at the Time of Radical Cystectomy (RC)
Description: Tumors will be assessed in a standard manner and given grade/stage according to the American Joint Commission on Cancer (AJCC) criteria. Efficacy will be assessed based on pathologic criteria and evidence of pharmacologic activity in the target tissue.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion
Number analyzed (Participants) | 8
Participants
  Complete pathological response | 2
  Pathologic downstaging | 4

2. Primary Outcome: Immunohistochemistry (IHC) Analyses of Pre-treatment (at TURBT) and Post-treatment (at Radical Cystectomy) Bladder Tumor Tissues Were Performed to Determine Whether Neoadjuvant Fosciclopirox Treatment Affected the Notch Cell Signaling Pathway.
Description: Immunohistochemistry (IHC) analyses of pre-treatment (at TURBT) and post-treatment (at radical cystectomy) bladder tumor tissues were performed to determine whether neoadjuvant fosciclopirox treatment affected the Notch cell signaling pathway. Immunohistochemistry staining intensity score as a measure of protein expression with four categories: negative (0), weak (1), moderate (2), and strong (3). Staining intensity scores were assigned by a blinded pathologist who specializes in genitourinary cancers. Pre-treatment and post-treatment bladder tumor samples were available for IHC analysis for six of the nine patients studied. For two patients, pre-treatment bladder tumor tissue samples obtained from TURBT at referring sites were not processed for IHC analysis. One patient was discovered to have metastatic MIBC after enrollment, and therefore, did not undergo RC, hence, no post-treatment sample was available for IHC analysis.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-treatment: CPX-POM, 900 mg/m^2 by 20-minute IV Infusion: Pre-treatment
- Post-treatment: CPX-POM, 900 mg/m^2 by 20-minute IV Infusion: Post-treatment
Arm/Group | Pre-treatment: CPX-POM, 900 mg/m^2 by 20-minute IV Infusion | Post-treatment: CPX-POM, 900 mg/m^2 by 20-minute IV Infusion
Number analyzed (Participants) | 6 | 6
score on a scale
  Notch 1 | 2.2 (0.8) | 1.3 (1.5)
  Notch 2 | 1.0 (0.9) | 0.2 (0.4)
  Notch 3 | 2.5 (1.2) | 1.5 (1.6)
  Jagged 1 | 2.0 (1.3) | 1.0 (1.5)
  Presenilin 1 | 1.3 (1.5) | 1.0 (1.3)
  Nicastrin | 2.5 (0.2) | 1.5 (1.6)
  Hes 1 | 1.5 (1.2) | 0.5 (1.2)
  Cyclin D1 | 0.0 (0.0) | 0.2 (0.4)
  CD8+ | 1.5 (0.5) | 0.5 (0.5)

3. Secondary Outcome: Number of Participant With Any Serious Adverse Events (SAEs) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE Version 4.03)
Description: Incidence of Serious Adverse Events in subjects receiving CPX-POM.
Time Frame: 56 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion
Number analyzed (Participants) | 9
Participants | 0

4. Secondary Outcome: Number of Participant With Any Adverse Events (AEs) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE Version 4.03)
Description: Incidence of Adverse Events in subjects receiving CPX-POM.
Time Frame: 56 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-POM, 900 mg/m^2 by 20 Minute IV Infusion (N=9)
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Epigastric Discomfort (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Gait disturbance (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Micturition urgency (Renal and urinary disorders) | 2
Bladder spasm (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
COVID-19 (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Penile burnnig sensation (Reproductive system and breast disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI and Sponsor plan to publish the data.

DOCUMENTS (2):
  • Study Protocol (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04608045/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT04608045/SAP_001.pdf